CLINICAL TRIAL: NCT02204605
Title: Video-based Consensus Opinion for Hand and Upper Extremity Problems
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator left the institution.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P000132
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Pain
Keywords: patients; puzzling; conditions
MeSH Terms: conditions — Pain; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Visits are not videotaped
- Videoed Patients (Experimental): Patients will have their visit videotaped.
  Interventions: Behavioral: Video-based Consensus Opinion

INTERVENTIONS:
Behavioral: Video-based Consensus Opinion
  Arms: Videoed Patients

SUMMARY:
The investigators would like to determine if there is a difference in patient satisfaction among patients who have puzzling pain conditions and receive one evaluation from their treating physician, and those that receive an evaluation from their treating physician and from a group of consulting physicians by video. The investigators expect to enroll 128 patients at Massachusetts General Hospital.

DETAILED DESCRIPTION:
Before visiting a specialist, patients have assumptions regarding diagnosis, etiology, prognosis, and preferred treatment for their condition. Naturally, some of these assumptions may be inaccurate or incomplete or there may be room for debate and disagreement even among specialists. We are looking for ways to make unexpected and indeterminate aspects of an illness less unsettling for patients. When the hand surgeon's advice doesn't ring true, the patient may lose confidence in that provider. Sometimes the interaction can feel disrespectful and even adversarial. We are curious whether patient's satisfaction with diagnosis, surgeon, and treatment plan would improve if they were able to get an opinion from many surgeons at once. One feasible way to do that would be to show an edited and anonymized video to a set of hand surgeons for their opinions on diagnosis and treatment.

Primary study question:

1. Among patients with initially puzzling pains, there is no difference in satisfaction with diagnosis between patients that receive a video based consensus opinion and those that receive routine care from a single hand surgeon controlling for psychological factors, demographics, and initial and final diagnosis.

   Secondary study questions:
2. Among patients with initially puzzling pains, there is no difference in pain intensity and disability one month after the initial visit between patient that receive a consensus diagnosis and those that receive routine care from a single surgeon.
3. There is no variation in diagnosis between observers (Observers are hand surgeons viewing the visit video and consulting on the diagnosis).

ELIGIBILITY:
Inclusion Criteria:

* All patients (>18 years) presenting to Dr. David Ring with painful conditions that are puzzling (A puzzling pain condition is defined as Dr. Ring being puzzled about what is causing the pain. Subject eligibility based on this criterion will be determined by Dr. Ring).
* English fluency and literacy
* Able to provide informed consent

Exclusion Criteria:

* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Likert Scale for Satisfaction | At enrollment
Likert Scale for Satisfaction | 4-6 weeks

SECONDARY OUTCOMES:
Patient Self-Efficacy Questionnaire (PSEQ-2) | At enrollment
Patient Self-Efficacy Questionnaire (PSEQ-2) | 4-6 weeks
Patient Health Questionnaire (PHQ-2) | at enrollment
Patient Health Questionnaire (PHQ-2) | 4-6 weeks
QuickDASH (Disabilities of the Arm, Shoulder, and Hand) | At enrollment
QuickDASH (Disabilities of the Arm, Shoulder, and Hand) | 4-6 weeks
Numerical Rating Scale for Pain | at enrollment
Numerical Rating Scale for Pain | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States